CLINICAL TRIAL: NCT04803396
Title: An Ascending Dose Tolerability Study and Pharmacokinetic Assessment in Healthy Male and Female Volunteers After Single & Multiple Oral Administration of DF2755A
Brief Title: Ascending Dose Tolerability Trial and PK Assessment in Healthy Volunteers After Single & Multiple Oral Intake of DF2755A
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor decided to not proceed from SAD to MAD to explore the possibility of further studying PD.
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BPS0115; 2016-003629-41 (EudraCT Number)
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-11

CONDITIONS: no Condition
Keywords: Healthy volunteers
MeSH Terms: interventions — DF2755A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study is a double blind study. The analytical centre as well as the Investigator and the team and the subjects were in blind conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo RS/PKS/PDS/SS (Placebo Comparator): Placebo was administered once a day (oad) as matching oral capsules. The administration took place at around 8:00 a.m with 200 mL of tap water, in sitting position, in fasting conditions.
  Interventions: Other: Placebo
- DF2755A 50 mg - RS/PKS/PDS/SS (Experimental): The experimental drug was administered once a day (oad) as one oral capsule of 50 mg.
  The administration took place at around 8:00 a.m with 200 mL of tap water, in sitting position, in fasting conditions.
  Interventions: Drug: DF2755A
- DF2755A 150 mg - RS/PKS/PDS/SS (Experimental): The experimental drug was administered once a day (oad) as oral capsules. The administration took place at around 8:00 a.m with 200 mL of tap water, in sitting position, in fasting conditions.
  Interventions: Drug: DF2755A
- DF2755A 300 mg - RS/PKS/PDS/SS (Experimental): The experimental drug was administered once a day (oad) as oral capsules. The administration took place at around 8:00 a.m with 200 mL of tap water, in sitting position, in fasting conditions.
  Interventions: Drug: DF2755A
- DF2755A 600 mg - RS/PKS/PDS/SS (Experimental): The experimental drug was administered once a day (oad) as oral capsules. The administration took place at around 8:00 a.m with 200 mL of tap water, in sitting position, in fasting conditions.
  Interventions: Drug: DF2755A

INTERVENTIONS:
Drug: DF2755A — DF2755A was planned to be administered in two different parts:
  Part A: Single oral dose administration on D1 according to the randomization (50, 150, 300 and 300 mg oad).
  Part B: was planned (100 mg bid, 200 mg bid or 300 mg bid) but not performed (repeated oral administration from Day 1 to Day 14).
  Other Names: allosteric inhibitor of CXCR1/2
  Arms: DF2755A 150 mg - RS/PKS/PDS/SS; DF2755A 300 mg - RS/PKS/PDS/SS; DF2755A 50 mg - RS/PKS/PDS/SS; DF2755A 600 mg - RS/PKS/PDS/SS
Other: Placebo — Single oral dose administration on D1
  Other Names: Matching placebo
  Arms: Placebo RS/PKS/PDS/SS

SUMMARY:
Primary objective:

•To evaluate the tolerability and safety of ascending single doses of DF2755A in healthy adult male and female volunteers.

Secondary Objectives:

* To determine the pharmacokinetics parameters of DF2755A
* To establish a dose concentration-response relationship over a wide range of doses in order to select a narrower range of dose and dosing regimen to be subsequently studied in patients after single administration
* To evaluate the effect of ascending single doses on the pharmacodynamics parameters
* To compare metabolites pathway in Human with the one observed in animals

Please note that the study has been closed after Part A (single ascending doses), so all the objectives were revised accordingly.

DETAILED DESCRIPTION:
The study was a phase I, single center, double-blind, placebo controlled, randomized, ascending single doses study in healthy male and female volunteers.

The design consisted of a double blind comparison of the test compound versus placebo in which the dose is increased in successive treatment periods.

The escalating dose had the aim of achieving enough safety information on an interval of doses possibly encompassing both the effective dose and the maximum tolerated dose (defined as the highest dose devoid of any clinical signs/symptoms). Practically, of the two Parts planned - part A and Part B - only the Part A took place.

The Part A consisted of single doses of 50 mg oad, 150 mg oad, 450 mg oad or 700 mg oad of DF2755A tested in healthy male and female volunteers who were hospitalized approximately for 4 days (D-1 morning to D4 morning).

The planned Part B should have consisted of repeated doses of 100 mg bid, 200 mg bid or 300 mg bid of DF2755A) but it was not performed. Hence, the study was terminated at the end of Part A and, consequently, both the methodology and the endpoints were revised accordingly.

ELIGIBILITY:
Inclusion Criteria:

* For eligibility into the trial, subjects had to meet all the following inclusion criteria:

  1. Healthy male subject, aged between 18 and 55 years inclusive;
  2. Healthy female subject infertile or in post menopause for at least two years, aged between 18 and 60 years inclusive;
  3. Body Mass Index (BMI) between 18.5 and 29.9 kg/m2 inclusive and weight ≤ 90kg;
  4. Considered as healthy after a comprehensive clinical assessment (detailed medical history and complete physical examination);
  5. Normal Blood Pressure (BP) and Heart Rate (HR) at the screening visit after 10 minutes in supine position:

     * 90 mmHg ≤ Systolic Blood Pressure (SBP) ≤ 140 mmHg or 150mmHg for subject > 45 years,
     * 50 mmHg ≤ Diastolic Blood Pressure (DBP) ≤ 90 mmHg,
     * 40 bpm ≤ HR ≤ 100 bpm, Or considered NCs by investigators;
  6. Smoker < 5cigarettes per day who stop totally during the study;
  7. Normal ECG recording on a 12-lead ECG at the screening visit:

     * 120 < PR < 210 ms,
     * QRS < 120 ms,
     * QTcf ≤ 430 ms for male and < 450 ms for female,
     * No sign of any trouble of sinusal automatism, Or considered NCs by investigators;
  8. Normal oral temperature;
  9. 36.3°C < oral body temperature < 37.5°C;
  10. Laboratory parameters within the normal range of the laboratory (haematological, blood chemistry tests, urinalysis). Individual values out of the normal range can be accepted if judged clinically non relevant by the Investigator;
  11. Normal dietary habits;
  12. Able to communicate well with the Investigator, understand and comply with the requirements of the study, and understand and sign a written informed consent prior to selection;
  13. Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

Exclusion Criteria:

1. Subject has had a clinically significant illness in the six weeks before screening in the opinion of the Investigator.
2. Subject has had a serious adverse reaction or significant hypersensitivity to any drug, has a known clinically significant allergy to anti-inflammatory drugs or chemically related compounds or has a clinically significant allergy to drugs, foods or other materials (in the opinion of the Investigator). However, subjects with mild hayfever may be included in the study.
3. Subject has used prescription medication in the 14 days prior to dosing or over-the-counter preparations for 7 days prior to dosing (including vitamin supplements and herbal remedies), with the exception of paracetamol which was allowed during the study (maximum 500 mg per administration, total daily dose maximum 2 grams).
4. Subject has a significant history of drug/solvent abuse or a positive drugs of abuse (DOA) test at any time during the study.
5. Subject has a history of alcohol abuse in the last 5 years or currently drinks in excess of 21 and 14 units per week for males and female, respectively, or has a positive alcohol breath test (ABT) at any time during the study.
6. Subject is not willing to refrain from caffeine/xanthine containing products in the 48 hours prior to admission to the clinical unit on Day -1 and for the duration of the residential period.
7. Subject who has a positive human immunodeficiency virus (HIV) screen, Hepatitis B screen or Hepatitis C screen.
8. Subject has donated blood or blood products (e.g., plasma or platelets) within the three months prior to screening.
9. Subject who is not suitable to participate in the study in the opinion of the Investigator;
10. Subject who has participated in any clinical study with an investigational drug/device within three months prior to the first day of dosing.
11. Subject who is in the exclusion period from another study.
12. Administrative or legal supervision.
13. Subject who would receive more than 4500 euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study. -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2019-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yves Donazzolo, MD, MSc, Principal Investigator — Eurofins Optimed
Locations (1):
- Eurofins Optimed, Gières, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 subjects were screened in this study. 32 subjects were included: 24 males and 8 females. All subjects completed the part A of the study.
Groups:
- Placebo: Placebo was administered once a day (oad) as matching oral capsules. The administration took place at around 8:00 a.m with 200 mL of tap water, in sitting position, in fasting conditions.
- 50 mg DF2755A: The experimental drug was administered once a day (oad) as one oral capsule of 50 mg.
  The administration took place at around 8:00 a.m with 200 mL of tap water, in sitting position, in fasting conditions.
  DF2755A: DF2755A was planned to be administered in two different parts:
  Part A: Single oral dose administration on D1 according to the randomization (50, 150, 300 and 300 mg oad).
  Part B: was planned (100 mg bid, 200 mg bid or 300 mg bid) not performed (repeated oral administration from Day 1 to Day 14).
  Hence, only part A of the study was accomplished.
- 150 mg DF2755A; 300 mg DF2755A; 600 mg DF2755A: The experimental drug was administered once a day (oad) as oral capsules. The administration took place at around 8:00 a.m with 200 mL of tap water, in sitting position, in fasting conditions.
  DF2755A: DF2755A was planned to be administered in two different parts:
  Part A: Single oral dose administration on D1 according to the randomization (50, 150, 300 and 300 mg oad).
  Part B: was planned (100 mg bid, 200 mg bid or 300 mg bid) not performed (repeated oral administration from Day 1 to Day 14).
  Hence, only part A of the study was accomplished.
Period: Overall Study
Arm/Group | Placebo | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Started | 8 | 6 | 6 | 6 | 6
Completed | 8 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Randomized set (RS) was defined as all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 6 | 6 | 6 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (11.9) | 46.3 (8.8) | 48.8 (7.8) | 45.8 (5.8) | 36.5 (13.3) | 44.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 1 | 1 | 1 | 8
  Male | 4 | 5 | 5 | 5 | 5 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 0 | 0 | 2
  White | 6 | 6 | 6 | 6 | 6 | 30
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 8 | 6 | 6 | 6 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events by Severity
Description: Adverse Event (AE), is defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment/product.
  Serious Adverse Event or Reaction, is any untoward medical occurrence, that:
  * Results in death;
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability or incapacity
  * an important medical event/reaction that may jeopardize the patient and require medical / surgical intervention to prevent one of the outcomes above.
  Any AE (including laboratory test abnormalities, intercurrent illnesses or injuries, and/or study procedures related AE) reported spontaneously by the subjects, or observed by the Investigator, was recorded according to the procedures in force at Eurofins Optimed.
Time Frame: Throughout the study, up to Day 4
Population: Safety set: defined as all included subjects having taken at least one dose of study drug.
Measure: Number; unit: events
Groups:
- Placebo: Placebo was administered once a day (oad) as matching oral capsules. The administration took place at around 8:00 a.m. with 200 mL of tap water, in sitting position, in fasting conditions.
  DF2755A: DF2755A was planned to be administered in two different parts:
  Part A: Single oral dose administration on D1 according to the randomization (50, 150, 300 and 600 mg oad).
  Part B: was planned (100 mg bid, 200 mg bid or 300 mg bid) not performed (repeated oral administration from Day 1 to Day 14).
  Hence, only part A of the study was accomplished.
- 50 mg DF2755A: The experimental drug was administered once a day (oad) as one oral capsule of 50 mg.
  The administration took place at around 8:00 a.m. with 200 mL of tap water, in sitting position, in fasting conditions.
  DF2755A: DF2755A was planned to be administered in two different parts:
  Part A: Single oral dose administration on D1 according to the randomization (50, 150, 300 and 600 mg oad).
  Part B: was planned (100 mg bid, 200 mg bid or 300 mg bid) not performed (repeated oral administration from Day 1 to Day 14).
  Hence, only part A of the study was accomplished.
- 150 mg DF2755A; 300 mg DF2755A; 600 mg DF2755A: The experimental drug was administered once a day (oad) as oral capsules. The administration took place at around 8:00 a.m. with 200 mL of tap water, in sitting position, in fasting conditions.
  DF2755A: DF2755A was planned to be administered in two different parts:
  Part A: Single oral dose administration on D1 according to the randomization (50, 150, 300 and 600 mg oad).
  Part B: was planned (100 mg bid, 200 mg bid or 300 mg bid) not performed (repeated oral administration from Day 1 to Day 14).
  Hence, only part A of the study was accomplished.
Arm/Group | Placebo | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
events
  Mild | 0 | 0 | 0 | 1 | 0
  Moderate | 2 | 3 | 0 | 1 | 0
  Severe | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Cmax of DF2755A
Description: Cmax is the observed maximum plasma concentration of a product.
Time Frame: Day 1 (0,5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16 h post-dose); Day 2 (24, 36, 40h post-dose); Day 3 (48, 60 h post-dose); Day 4 (72 h post dose)
Population: The pharmacokinetic set (PKS) was defined as all the included subjects who have taken at least one dose of study drug without major protocol deviations affecting pharmacokinetics and with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 50 mg DF2755A: The experimental drug was administered once a day (oad) as one oral capsule of 50 mg.
  The administration took place at around 8:00 a.m. with 200 mL of tap water, in sitting position, in fasting conditions.
  DF2755A: DF2755A was planned to be administered in two different parts:
  Part A: Single oral dose administration on D1 according to the randomization (50, 150, 300 and 300 mg oad).
  Part B: was planned (100 mg bid, 200 mg bid or 600 mg bid) not performed (repeated oral administration from Day 1 to Day 14).
  Hence, only part A of the study was accomplished.
Arm/Group | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 1943 (39.0) | 6324 (28.7) | 16081 (20.2) | 26145 (32.0)

3. Secondary Outcome: Tmax
Description: It is the first time to reach Cmax.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 6 | 6 | 6 | 6
Hours | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.53] | 0.77 [0.50 to 3.00]

4. Secondary Outcome: t1/2
Description: It is the plasma concentration half life.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 6 | 5 | 5 | 5
Hours | 1.49 (54.2) | 1.62 (42.6) | 3.19 (43.9) | 4.05 (52.5)

5. Secondary Outcome: AUC0-t
Description: The area under the concentration vs. time curve from time zero (pre-dose) to the time of last quantifiable concentration was calculated using a linear trapezoidal method.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*ng/mL | 3314.54 (38.9) | 9498.72 (30.2) | 25354.16 (12.2) | 75915.63 (26.9)

6. Secondary Outcome: AUC 0-inf
Description: It is the area under the plasma concentration-time curve from administration up to infinity with extrapolation of the terminal phase.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 4 | 5 | 5 | 5
h*ng/mL | 4005.92 (39.7) | 9126.11 (13.2) | 26102.10 (13.8) | 81580.67 (26.4)

7. Secondary Outcome: Vz/F
Description: It is the apparent volume of distribution during terminal phase after non-intravenous administration.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Groups:
- 150 mg DF2755A: The experimental drug was administered once a day (oad) as oral capsules. The administration took place at around 8:00 a.m with 200 mL of tap water, in sitting position, in fasting conditions.
  DF2755A: DF2755A was planned to be administered in two different parts:
  Part A: Single oral dose administration on D1 according to the randomization (50, 150, 300 and 600 mg oad).
  Part B: was planned (100 mg bid, 200 mg bid or 300 mg bid) not performed (repeated oral administration from Day 1 to Day 14).
  Hence, only part A of the study was accomplished.
Arm/Group | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 6 | 5 | 5 | 5
liters | 27.74 (48.6) | 38.33 (32.7) | 52.98 (36.1) | 42.98 (31.2)

8. Secondary Outcome: CL/F
Description: It is the apparent oral clearance of the drug, where CL = clearance and F = bioavailability.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hours
Arm/Group | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 6 | 5 | 5 | 5
L/hours | 12.87 (31.2) | 16.44 (14.5) | 11.49 (13.4) | 7.35 (27.7)

9. Secondary Outcome: Ae,f(0-72) Total Amount in Faeces
Description: After oral administration, the individual amount of the drug excreted in faeces as DF2755Y is measured by the tracing of the radiolabelled compound [14C]DF2755A.
Time Frame: 0-24 h post-dose; 24-48 h post-dose, 48-72 h post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg
Arm/Group | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 4 | 5 | 5 | 6
μg | 50.04 (81.2) | 220.92 (78.5) | 425.62 (61.1) | 316.38 (83)

10. Secondary Outcome: Fe,f(0-72)
Description: The individual corresponding fraction of DF2755A dose excreted in faeces as DF2755Y over time in the whole sampling window is reported.
Time Frame: 0-24 h post-dose; 24-48 h post-dose, 48-72 h post dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of value
Groups:
- 50 mg DF2755A: The experimental drug was administered once a day (oad) as one oral capsule of 50 mg.
  The administration took place at around 8:00 a.m with 200 mL of tap water, in sitting position, in fasting conditions.
  DF2755A: DF2755A was planned to be administered in two different parts:
  Part A: Single oral dose administration on D1 according to the randomization (50, 150, 300 and 600 mg oad).
  Part B: was planned (100 mg bid, 200 mg bid or 300 mg bid) not performed (repeated oral administration from Day 1 to Day 14).
  Hence, only part A of the study was accomplished.
- 300 mg DF2755A: The experimental drug was administered once a day (oad) as oral capsules. The administration took place at around 8:00 a.m with 200 mL of tap water, in sitting position, in fasting conditions.
  DF2755A: DF2755A was planned to be administered in two different parts:
  Part A: Single oral dose administration on D1 according to the randomization (50, 150, 300 and 300 mg oad).
  Part B: was planned (100 mg bid, 200 mg bid or 600 mg bid) not performed (repeated oral administration from Day 1 to Day 14).
  Hence, only part A of the study was accomplished.
- 600 mg DF2755A: The experimental drug was administered once a day (oad) as oral capsules. The administration took place at around 8:00 a.m with 200 mL of tap water, in sitting position, in fasting conditions.
  DF2755A: DF2755A was planned to be administered in two different parts:
  Part A: Single oral dose administration on D1 according to the randomization (50, 150, 300 and 600 mg oad).
  Part B: was planned (100 mg bid, 200 mg bid or 300 mg bid) not performed (repeated oral administration from Day 1 to Day 14).
  Hence, only part A of the study was accomplished.
Arm/Group | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 4 | 5 | 5 | 6
percentage of value | 0.11 (81.2) | 0.17 (78.5) | 0.16 (61.1) | 0.06 (83)

11. Secondary Outcome: Ae,ur(0-72)
Description: The individual amount of DF2755A excreted in urine as DF2755Y over time in the whole sampling window is reported.
Time Frame: 0-6 h post-dose; 6-10 h post-dose; 10-16h post-dose; 16-24h post-dose; 24-48h post-dose; 48-72h post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg
Groups:
- 300 mg DF2755A; 600 mg DF2755A: The experimental drug was administered once a day (oad) as oral capsules. The administration took place at around 8:00 a.m with 200 mL of tap water, in sitting position, in fasting conditions.
  DF2755A: DF2755A was planned to be administered in two different parts:
  Part A: Single oral dose administration on D1 according to the randomization (50, 150, 300 and 600 mg oad).
  Part B: was planned (100 mg bid, 200 mg bid or 300 mg bid) not performed (repeated oral administration from Day 1 to Day 14).
  Hence, only part A of the study was accomplished.
Arm/Group | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 6 | 6 | 6 | 6
μg | 3612.8 (32.7) | 3556.2 (38.1) | 12110.41 (74.1) | 20018.07 (27)

12. Secondary Outcome: Fe,ur(0-72)
Description: The individual corresponding fraction of DF2755A dose excreted in urine as DF2755Y over time in the whole sampling window is reported.
Time Frame: 0-6 h post-dose; 6-10 h post-dose; 10-16h post-dose; 16-24h post-dose; 24-48h post-dose; 48-72h post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of value
Arm/Group | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage of value | 8.14 (32.7) | 2.67 (38.1) | 4.55 (74.1) | 3.76 (27)

13. Secondary Outcome: CLR
Description: It is the renal clearance of DF2755Y.
Time Frame: 0-6 h post-dose; 6-10 h post-dose; 10-16h post-dose; 16-24h post-dose; 24-48h post-dose; 48-72h post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hours
Arm/Group | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 6 | 6 | 6 | 6
L/hours | 1.09 (34) | 0.37 (50.4) | 0.48 (70.1) | 0.26 (27.8)

14. Secondary Outcome: 12-lead ECG (HR)
Description: 12-lead ECG included the assessment of the following parameters: HR, PR, QRS, QT, and QTcF. Here heart rate (HR) is reported. Heart rate (or pulse rate is the frequency of the heartbeat measured by the number of contractions (beats) of the heart per minute (bpm). The heart rate can vary according to the body's physical needs, including the need to absorb oxygen and excrete carbon dioxide, but is also modulated by numerous factors, including, but not limited to, genetics, physical fitness, stress or psychological status, diet, drugs, hormonal status, environment, and disease/illness as well as the interaction between and among these factors. It is usually equal or close to the pulse measured at any peripheral point.
Time Frame: day -1 (pre treatment), day 3 (last visit after treatment)
Population: The Safety set (SS) was defined as all included subjects having taken at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: bpm
Groups:
- Placebo RS/PKS/PDS/SS: Placebo was administered once a day (oad) as matching oral capsules. The administration took place at around 8:00 a.m. with 200 mL of tap water, in sitting position, in fasting conditions.
  Placebo: Single oral dose administration on D1
- DF2755A 50 mg - RS/PKS/PDS/SS: The experimental drug was administered once a day (oad) as one oral capsule of 50 mg.
  The administration took place at around 8:00 a.m. with 200 mL of tap water, in sitting position, in fasting conditions.
  DF2755A: DF2755A was planned to be administered in two different parts:
  Part A: Single oral dose administration on D1 according to the randomization (50, 150, 300 and 600 mg oad).
  Part B: was planned (100 mg bid, 200 mg bid or 300 mg bid) but not performed (repeated oral administration from Day 1 to Day 14).
- DF2755A 150 mg - RS/PKS/PDS/SS; DF2755A 300 mg - RS/PKS/PDS/SS: The experimental drug was administered once a day (oad) as oral capsules. The administration took place at around 8:00 a.m. with 200 mL of tap water, in sitting position, in fasting conditions.
  DF2755A: DF2755A was planned to be administered in two different parts:
  Part A: Single oral dose administration on D1 according to the randomization (50, 150, 300 and 600 mg oad).
  Part B: was planned (100 mg bid, 200 mg bid or 300 mg bid) but not performed (repeated oral administration from Day 1 to Day 14).
- DF2755A 600 mg - RS/PKS/PDS/SS: The experimental drug was administered once a day (oad) as oral capsules. The administration took place at around 8:00 a.m with 200 mL of tap water, in sitting position, in fasting conditions.
  DF2755A: DF2755A was planned to be administered in two different parts:
  Part A: Single oral dose administration on D1 according to the randomization (50, 150, 300 and 600 mg oad).
  Part B: was planned (100 mg bid, 200 mg bid or 300 mg bid) but not performed (repeated oral administration from Day 1 to Day 14).
Arm/Group | Placebo RS/PKS/PDS/SS | DF2755A 50 mg - RS/PKS/PDS/SS | DF2755A 150 mg - RS/PKS/PDS/SS | DF2755A 300 mg - RS/PKS/PDS/SS | DF2755A 600 mg - RS/PKS/PDS/SS
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
bpm
  D-1 | 67.8 (10.7) | 66.7 (6.3) | 59.3 (4.4) | 65.2 (7.4) | 60.7 (12.7)
  D3 | 61.3 (8.3) | 58.2 (4.4) | 55.0 (6.4) | 62.2 (4.6) | 58.8 (12.4)

15. Secondary Outcome: 12-lead ECG PR, QRS, QT, and QTcF
Description: It included the assessment of the following parameters: PR, QRS, QT, and QTcF. PR=PR interval measured on ECG; it is the period, measured in milliseconds, that extends from the beginning of the P wave (the onset of atrial depolarization) until the beginning of the QRS complex (the onset of ventricular depolarization).
  QRS=QRS interval measured on ECG; It's the combination of 3 of the graphical deflections seen on a typical ECG. It corresponds to the depolarization of the right and left ventricles of the heart and contraction of the large ventricular muscles.
  QT=QT interval; it is used to assess some of the electrical heart properties, calculated as the time from the start of the Q wave to the end of the T wave, and approximates to the time taken from when the cardiac ventricles start to contract to when they finish relaxing.
  QtcF=QT interval corrected for heart rate using Fridericia's formula; it's measured with a "QT/QTcF semiautomated triplicate averaging method" (TAM).
Time Frame: day -1 (pre treatment), day 3 (last visit after treatment)
Population: The Safety set (SS) was defined as all included subjects having taken at least one dose of study drug
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Placebo: Placebo was administered once a day (oad) as matching oral capsules. The administration took place at around 8:00 a.m. with 200 mL of tap water, in sitting position, in fasting conditions.
Arm/Group | Placebo | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
ms
  PR D-1 | 164.3 (19.7) | 187.0 (14.7) | 166.3 (15.5) | 156.7 (20.7) | 160.3 (27.6)
  PR D3 | 167.3 (18.1) | 192.7 (15.9) | 170.3 (24.8) | 166.0 (19.8) | 162.3 (20.6)
  QRS D-1 | 85.8 (8.3) | 87.7 (9.1) | 90.0 (8.2) | 88.3 (15.6) | 91.3 (13.7)
  QRS D3 | 83.5 (8.8) | 82.7 (5.0) | 87.7 (9.4) | 87.3 (13.0) | 90.0 (12.8)
  QT D-1 | 383.5 (35.7) | 380.7 (10.5) | 390.3 (24.1) | 399.7 (23.3) | 397.3 (27.4)
  QT D3 | 394.5 (33.6) | 386.3 (12.1) | 404.0 (21.1) | 401.3 (16.0) | 400.7 (29.4)
  QTcF D-1 | 397.1 (26.7) | 394.0 (8.6) | 388.0 (17.7) | 410.2 (18.2) | 400.2 (25.7)
  QTcF D3 | 395.9 (27.5) | 381.5 (11.3) | 391.5 (15.5) | 406.0 (13.2) | 395.0 (14.0)

16. Secondary Outcome: Systolic and Diastolic Blood Pressure (SBP, DBP)
Description: Vital signs included SBP and DBP in both supine position (after 10 minutes rest) and standing position (after 2 minutes).
  SBP= Systolic Blood Pressure is the maximum pressure during one heartbeat. DBP= Diastolic Blood Pressure minimum is the pressure between two heartbeats.
Time Frame: day -1 (pre treatment), day 2 (post-treatment)
Population: The Safety set (SS) was defined as all included subjects having taken at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
mmHg
  Supine SBP D-1 | 110.4 (13.7) | 112.2 (11.5) | 114.2 (14.1) | 108.2 (6.7) | 113.8 (8.8)
  Supine SBP D2 | 110.8 (9.8) | 106.0 (6.8) | 113.0 (15.9) | 102.8 (12.1) | 104.8 (5.0)
  Standing SBP D-1 | 111.6 (12.6) | 116.3 (16.5) | 120.5 (8.7) | 115.7 (9.5) | 115.2 (2.6)
  Standing SBP D2 | 107.0 (14.4) | 101.8 (12.0) | 118.2 (15.9) | 111.2 (13.2) | 112.7 (11.8)
  Supine DBP D-1 | 65.3 (7.6) | 64.7 (3.3) | 65.0 (5.2) | 64.7 (8.9) | 61.0 (6.7)
  Supine DBP D2 | 64.3 (6.2) | 63.5 (2.6) | 69.8 (9.4) | 64.5 (11.7) | 63.3 (6.0)
  Standing DBP D-1 | 75.8 (5.6) | 72.2 (7.2) | 74.0 (4.4) | 72.7 (11.6) | 78.7 (7.0)
  Standing DBP D2 | 74.0 (5.5) | 71.7 (5.4) | 77.3 (8.0) | 72.0 (9.9) | 73.3 (7.3)

17. Secondary Outcome: Heart Rate (HR)
Description: Vital signs included HR in both supine position (after 10 minutes rest) and standing position (after 2 minutes).
  HR: Heart Rate(or pulse rate) is the frequency of the heartbeat measured by the number of contractions (beats) of the heart per minute (bpm).
Time Frame: day -1 (pre treatment), day 3 (last visit after treatment)
Population: The Safety set (SS) was defined as all included subjects having taken at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
bpm
  Supine HR D-1 | 65.8 (6.5) | 63.3 (5.9) | 63.3 (4.7) | 65.3 (8.7) | 57.3 (7.8)
  Supine HR D3 | 64.0 (6.5) | 61.3 (5.3) | 63.3 (4.7) | 56.3 (6.3) | 58.2 (11.2)
  Standing HR D-1 | 76.3 (7.9) | 74.3 (3.2) | 76.7 (6.8) | 69.5 (11.1) | 70.7 (10.6)
  Standing HR D3 | 73.6 (5.9) | 74.0 (11.0) | 70.3 (8.0) | 66.7 (6.7) | 72.8 (10.2)

18. Secondary Outcome: Oral Body Temperature
Description: The oral body temperature is the measurement of the body temperature placing the thermometer under one side of the back of the tongue. Human body temperature varies. It depends on sex, age, time of day, exertion level, health status (such as illness and menstruation), what part of the body the measurement is taken at, state of consciousness (waking, sleeping, sedated), and emotions. Body temperature range in this study was 36.3 to 37.5 °C.
Time Frame: day -1 (pre treatment), day 2 (post-treatment)
Population: The Safety set (SS) was defined as all included subjects having taken at least one dose of study drug
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Placebo | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
°C
  Oral Temperature D-1 | 36.41 (0.24) | 36.32 (0.20) | 36.38 (0.13) | 36.40 (0.23) | 36.32 (0.37)
  Oral Temperature D2 | 36.38 (0.27) | 36.40 (0.14) | 36.30 (0.30) | 36.28 (0.23) | 36.13 (0.27)

ADVERSE EVENTS:
Time Frame: adverse event data were collected from baseline (day -21) up to end of study visit (day 4)
Description: All subjects who received a dose of the study drug were included in the safety evaluation (Safety Set N=32).
Groups:
- Placebo: Placebo was administered once a day (oad) as matching oral capsules. The administration took place at around 8:00 a.m with 200 mL of tap water, in sitting position, in fasting conditions.
  Hence, only part A of the study was accomplished.
Arm/Group | Placebo | 50 mg DF2755A | 150 mg DF2755A | 300 mg DF2755A | 600 mg DF2755A
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/8 | 1/6 | 0/6 | 1/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | 50 mg DF2755A (N=6) | 150 mg DF2755A (N=6) | 300 mg DF2755A (N=6) | 600 mg DF2755A (N=6)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of subjects analysed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT04803396/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT04803396/SAP_001.pdf